CLINICAL TRIAL: NCT06427239
Title: A Single-center, Open-label, Exploratory Study of HRS-4642 Combined With Adebelimab in the Treatment of Advanced Pancreatic Cancer
Brief Title: Exploratory Clinical Study of HRS-4642 Combined With Adebelimab in the Treatment of Advanced Pancreatic Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Xian-Jun Yu, Professor, Fudan University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PANC-2nd-IIT-HRS4642-SHR1316
Record Dates: First submitted 2024-05-19; First posted 2024-05-23 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dose Escalation 300mg (Experimental): For HRS-4642 in combination with Adebrelimab, for advanced or metastatic pancreatic ductal adenocarcinoma.
  Interventions: Drug: HRS-4642; Drug: Adebrelimab
- Dose Escalation 400mg (Experimental): For HRS-4642 in combination with Adebrelimab, for advanced or metastatic pancreatic ductal adenocarcinoma.
  Interventions: Drug: HRS-4642; Drug: Adebrelimab
- Dose Escalation 500mg (Experimental): For HRS-4642 in combination with Adebrelimab, for advanced or metastatic pancreatic ductal adenocarcinoma.
  Interventions: Drug: HRS-4642; Drug: Adebrelimab

INTERVENTIONS:
Drug: HRS-4642 — HRS-4642 will be administrated per dose level in which the patients are assigned.
Drug: Adebrelimab — Adebrelimab will be administrated per dose level in which the patients are assigned

SUMMARY:
The study is being conducted to evaluate the safety, tolerability and efficacy of HRS-4642 combined with adebelimab in subjects with locally advanced or metastatic pancreatic ductal adenocarcinoma.

DETAILED DESCRIPTION:
This study is an open, single center, exploratory clinical trial aimed at evaluating the efficacy and safety of HRS-4642 combined with adebelimab in the treatment of patients with unresectable locally advanced or metastatic pancreatic ductal adenocarcinoma.

This study experiment is divided into two stages: dose exploration stage and efficacy exploration stage. During the dose exploration phase, RP2D was determined based on the safety, tolerability, and preliminary efficacy data of HRS-4642 combined with adelbizumab treatment, and then entered the efficacy exploration phase.

ELIGIBILITY:
Inclusion Criteria:

1. Patients volunteered to participate in this study and signed informed consent;
2. Age: ≥18 and ≤75 years old, male or female;
3. Advanced (metastatic or unresectable) Pancreatic ductal adenocarcinoma; and subjects must have at least one measurable lesion as defined by RECIST v1.1;
4. With failure or absence of standard treatment, and progress within 6 months of adjuvant therapy can also be included in the study;
5. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1;
6. Life expectancy ≥ 12 weeks;
7. Adequate marrow and organ function;
8. AE caused by previous anti-tumor therapy must be restored to ≤ level 1 (CTCAE v5.0) or a stable state evaluated by the researcher, except for hair loss (any level) and peripheral neuropathy of level 2;
9. Female participants of childbearing age must undergo a pregnancy test within one week before the start of the study medication, and the result is negative. They are willing to use a medically recognized and efficient contraceptive method during the study period and within three months after the last administration of the study medication; For male participants whose partners are women of childbearing age, they should agree to use effective methods of contraception during the study period and within 3 months after the last study administration;

Exclusion Criteria:

1. Known to be allergic to the investigational drug or any of its components;
2. Have other active malignancies within 5 years;
3. Systemic antitumor therapy was received 4 weeks before the start of the study, and palliative radiotherapy was completed within 14 days before the first dose;
4. Previously received allogeneic hematopoietic stem cell transplantation or organ transplantation;
5. Accompanied by untreated or active central nervous system (CNS) metastases;
6. Within 6 months prior to entering the study, patients with severe cardiovascular and cerebrovascular thromboembolism;
7. Hypertension with poor drug control (continuous increase in systolic blood pressure ≥ 150mm Hg or diastolic blood pressure ≥ 100mmHg);
8. Late stage patients with symptoms that have spread to the internal organs and are at risk of life-threatening complications in the short term;
9. With interstitial lung disease, non-infectious pneumonia, severe and uncontrolled internal medicine diseases, acute infections, recent history of major surgery (within 28 days or not yet recovered from side effects);
10. Participated in clinical trials of any drug or medical device within 4 weeks prior to the first administration;
11. With congenital or acquired immune deficiency, such as people infected with HIV, active hepatitis B (HBV DNA ≥ 500 IU/ml), hepatitis C (hepatitis C antibody positive, and HCV-RNA higher than the detection limit of the analytical method) or combined with hepatitis B and hepatitis C infection;
12. With any active autoimmune diseases or a history of autoimmune diseases;
13. Received systemic treatment with corticosteroids or other immunosuppressants within 2 weeks prior to the first medication;
14. High risk of pancreatitis, serum amylase and/or lipase concentrations ≥ 3 times ULN; who have a simple increase in lipase, will be considered for inclusion by the researchers;
15. Other situations that researchers believe should not be included.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-05-29 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Dose Limited Toxicity (DLT) | Day 1 to Day 21 after the first combination therapy was administrated
  A DLT is defined as any event meeting the DLT criteria occurring within 21 days of first dose on Cycle 1 Day 1 (C1D1), excluding toxicities clearly related to disease progression or intercurrent illness
Recommended phase II dose (RP2D) | Approximately 12 months
  RP2D will be determined on the basis of evaluation on safety and efficacy data in dose escalation stages.
Objective Response Rate (ORR) | Up to approximately 12 months
  Evaluated by RECIST v1.1.

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | Up to approximately 12 months
  Evaluated by RECIST v1.1.
Duration of Response (DOR) | Up to approximately 12 months
  Evaluated by RECIST v1.1.
Progression Free Survival (PFS) | Up to approximately 12 months
  Time from the date of enrollment to of disease progression, or death of any cause, or date of lost follow-up, whichever comes first, otherwise subject data were censored at time last known disease free.
Overall survival (OS) | Up to approximately 12 months
  Time from the date of enrollment to data of death from any cause, or date of lost follow-up, whichever comes first, and otherwise censored at time last known alive.
Adverse events (AEs) | From the first drug administration to within 90 days for the last adebrelimab dose
  AEs are assessed by NCI-CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Pancreatic Surgery, Fudan University Shanghai Cancer Center; Pancreatic Cancer Institute, Fudan University, Shanghai, Shanghai Municipality, China